CLINICAL TRIAL: NCT02843503
Title: Factors in Accuracy Studies Influencing Measured CGM Performance: a Comparison of Measured Continuous Glucose Monitor Performance Using Venous, Arterialized-venous and Capillary Reference Glucose Samples.
Brief Title: Factors in Accuracy Studies Influencing Measured CGM Performance.
Acronym: FACT-CGM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, J.H. DeVries, professor of diabetes medicine, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL57491.018.16
Record Dates: First submitted 2016-07-19; First posted 2016-07-26 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arterialized-venous reference YSI (Experimental): CGM monitoring performance per arterialized venous reference measurement (YSI)
  Interventions: Device: Arterialized-venous reference (YSI)
- Venous reference samples YSI (Experimental): CGM monitoring performance per venous reference measurement (YSI)
  Interventions: Device: Venous reference measurement (YSI); Device: Capillary reference (SMBG)

INTERVENTIONS:
Device: Arterialized-venous reference (YSI) — All patients will be fitted with the a CGM system, Dexcom G5 Mobile, patients receive an iv-catheter to sample venous blood. The samples will be arterialized using a heated-hand-box (arterialized-venous reference (YSI). Blood will be drawn for the determination of glucose concentrations using arterialized-venous sampling techniques per YSI.
  Arms: Arterialized-venous reference YSI
Device: Venous reference measurement (YSI) — All patients will be fitted with the a CGM system, Dexcom G5 Mobile, patients receive an iv-catheter to sample venous blood. Blood will be drawn for the determination of glucose concentrations using venous sampling techniques measured per YSI.
  Arms: Venous reference samples YSI
Device: Capillary reference (SMBG) — All patients will be fitted with the a CGM system, Dexcom G5 Mobile, patients receive vingerstick measurements to sample capillary blood measured per Self Monitoring of Blood Glucose (SMBG) device.
  Arms: Venous reference samples YSI

SUMMARY:
Primary objective is to assess the impact of different reference glucose measurement methods on the measured performance of a CGM system, aiming at further standardization for the assessment of CGM systems. Secondary objective is to describe the relationship between glucose concentration of venous, capillary and arterialized-venous measurement samples.

Study design: Open-label trial. Study population: Nineteen patients with type 1 diabetes aged 18 years and older will be included.

Intervention: The study will use the Dexcom G5 Mobile CGM. The participant will visit the clinical research center (CRC) twice during a 6 day period. These visits will have a duration of 8 hours. Blood will be drawn for the determination of glucose concentrations using venous, arterialized-venous and capillary sampling techniques. The patient will receive his usual breakfast and an increased insulin bolus will be administered to correct the breakfast glucose excursion with the aim of inducing a period of minor hypoglycemia. Blood sampling will continue until the end of the admission. The sensor will be worn until the end of the second 8-hour CRC session, which will be planned on day 6 or earlier depending on patient preference. The sensor will be removed and their sensor and blood glucose meter data downloaded from the devices. In the case of sensor failure before the first CRC session, patients will be instructed to insert a new sensor per the manufacturer's instruction and to notify study staff of the event. In case of failure of the sensor after the first CRC session but before the second CRC session, patients will return to the CRC for sensor removal and for data download.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with type 1 DM at least 6 months according to the WHO definition
* Body Mass Index (BMI) <35 kg/m²
* willing and able to wear a CGM device for the duration of the study and undergo all study procedures
* HbA1c <10%
* Signed informed consent form prior to study entry

Exclusion Criteria:

* patient is pregnant, or breast feeding during the period of the study.
* patient is using a medication that significantly impacts glucose metabolism (oral steroids) except if stable for at least the last three months and expected to remain stable for the study duration.
* patient requires regular use of acetaminophen (paracetamol) while participating in the study due to known negative impact on CGM performance.
* patient is actively enrolled in another clinical trial or took part in a study within 30 days.
* known adrenal gland problem, panhypopitutarism, gastroparesis, migraine, epilepsy or ischemic heart disease or other cardiovascular event in the year previous to study participation .
* inability of the patient to comply with all study procedures.
* inability of the patient to understand the patient information.
* patient donated blood in the last 3 months.
* has severe medical or psychological condition(s) or chronic conditions/infections that in the opinion of the investigator would compromise the patient's safety or successful participation in the study.
* is assessed by the investigators to have difficult intravenous (IV) access .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Mean Absolute Relative Difference (MARD) | up to day 6 of use
  MARD will be assessed per average of the 8 hour arterialization and regular venous study visit.

SECONDARY OUTCOMES:
Accuracy of sensors (MARD) per hypoglycemic range | up to day 6 of use
  Accuracy of the sensor in the hypoglycaemic (defined as a blood glucose value ≤70 mg/dL) area as an average of the first six days of use.
Accuracy (MARD) of sensors per hyperglycemic range | up to day 6 of use
  Accuracy of the sensor in the hyperglycaemic (defined as a blood glucose value >180 mg/dL) area as an average of the first six days of use.
Glucose content (mg/dL) of venous reference samples. | Up day 6 of study during both intervention visits
  Glucose content of venous reference samples will be measured per YSI.
Glucose content (mg/dL) of venous-arterialized reference samples. | up day 6 of study during both intervention visits
  Glucose content of venous-arterialized reference samples will be measured per YSI.
Glucose content (mg/dL) of capillary reference samples. | up day 6 of study during both intervention visits
  Glucose content of capillary reference samples will be measured per SMBG.

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No